CLINICAL TRIAL: NCT01147692
Title: An Open-label, Sequential Study to Evaluate the Pharmacokinetics of Simvastatin When Coadministered With Albiglutide in Healthy Adult Subjects
Brief Title: A Drug Interaction Study of Simvastatin and Albiglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 108366
Record Dates: First submitted 2010-04-29; First posted 2010-06-22 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: albiglutide; simvastatin; healthy volunteers; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Simvastatin; rGLP-1 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- simvastatin plus albiglutide (Experimental): A single dose of 80mg simvastatin on Day 1 followed by 5 weekly doses of subcutaneous albiglutide followed by a single dose of 80mg simvastatin on Day 38.
  Interventions: Biological: simvastatin plus albiglutide

INTERVENTIONS:
Biological: simvastatin plus albiglutide — A single dose of 80mg simvastatin on Day 1 followed by 5 weekly doses of subcutaneous albiglutide followed by a single dose of 80mg simvastatin on Day 38.

SUMMARY:
This open-label study evaluates the pharmacokinetics of simvastatin when coadministered with albiglutide in healthy adult subjects. The primary objective is to assess the effect of albiglutide doses on the pharmacokinetics of simvastatin.

DETAILED DESCRIPTION:
This Phase I open-label study evaluates the pharmacokinetics of simvastatin when coadministered with albiglutide in healthy adult subjects. The primary objective is to assess the effect of albiglutide doses on the pharmacokinetics of simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* no clinically significant diseases or clinically significant abnormal laboratory values
* females must be of non-childbearing potential
* body mass index (BMI) is >/=18 kg and ≤30 kg/m2
* nonsmoker
* negative drug screen

Exclusion Criteria:

* positive test results for hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
* any clinically relevant abnormality
* female subject is pregnant or breast-feeding
* history of any anaphylactic reaction to any drug
* history of significant cardiovascular or pulmonary dysfunction
* current or chronic history of liver disease
* history of alcohol or substance abuse
* history of thyroid dysfunction or disease
* history of gastrointestinal surgery or disease
* history of pancreatitis
* previously received any GLP-1 mimetic compound (e.g., exenatide)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2010-08-27 (Actual); Study Completion 2010-08-27 (Actual)

PRIMARY OUTCOMES:
The effect of albiglutide on the pharmacokinetics of simvastatin | 42 days

SECONDARY OUTCOMES:
The pertinent plasma pharmacokinetic parameters of simvastatin with and without albiglutide | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Young MA, Wald JA, Matthews JE, Scott R, Hodge RJ, Zhi H, Reinhardt RR. Clinical pharmacology of albiglutide, a GLP-1 receptor agonist. Postgrad Med. 2014 Nov;126(7):84-97. doi: 10.3810/pgm.2014.11.2836. PMID 25387217
- See also: Results for study 108366 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/108366?search=study&study_ids=108366#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 108366 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108366 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108366 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108366 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108366 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108366 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108366 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register